CLINICAL TRIAL: NCT05265598
Title: Is This PJI Really Acute: A Quantitative Sonication Fluid Analysis
Brief Title: Is This PJI Really Acute: A Quantitative Sonication Fluid Analysis (Sonic)
Acronym: Sonic
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01113; mu22Clauss
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Prosthetic-joint Infection
Keywords: debridement, antibiotics and implant retention (DAIR); sonication fluid analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective study is to analyse microbiological cultures from the sonication fluid of the explanted prothesis to detect bacteria in the biofilm on the implant surface and to investigate whether the number of bacteria in the biofilm correlates with the duration of the PJI respectively with the period between symptom onset and date of revision surgery.

DETAILED DESCRIPTION:
Implant associated infections in orthopaedics and trauma surgery are a well-known and feared complication. Prosthetic-joint infection (PJI) is caused by a biofilm which is located atop the surface of the implant which as growing with the duration of the PJI. This retrospective study is to analyse microbiological cultures from the sonication fluid of the explanted prothesis to detect bacteria in the biofilm on the implant surface and to investigate whether the number of bacteria in the biofilm correlates with the duration of the PJI respectively with the period between symptom onset and date of revision surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent a revision surgery of hip, knee and shoulder arthroplasties operated at the university hospital of Basel between 2011 and 2021,
* patients who had a PJI as a suspected diagnosis and
* have microbiological cultures from sonication fluid from removed prosthesis.

Exclusion Criteria:

* patients in the database who

  1. have non-bacterial microbiological positive cultures (e.g. fungal infection) and
  2. have not received a sonication of the removed prosthesis during the diagnostic process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the required criteria will be extracted from an existing clinical consultation database of the clinic of infectious disease. All patients in this database were treated and recorded on a consultative base between 2011 and 2021 by the Department of Orthopaedics and Traumatology and the Department of Infectious Diseases at the University Hospital Basel for a suspected PJI.
Sampling Method: Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-03-11 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
number of bacteria | one time assessment at baseline
  number of bacteria detected during revision surgery will be taken from the sonication fluid and the quantitative analysis of the microbiological samples
duration of the infection | one time assessment at baseline
  duration of the infection

CONTACTS AND LOCATIONS:
Overall Officials: Martin Clauss, PD Dr. med., Principal Investigator — Department of Orthopaedics and Traumatology, University Hospital Basel
Locations (1):
- Department of Orthopaedics and Traumatology, University Hospital Basel, Basel, Switzerland